CLINICAL TRIAL: NCT03951636
Title: Non Surgical Protocol for Treatment of Mucositis Using an Er:YAG Laser or an Air-abrasive Device: a Randomized Clinical Trial
Brief Title: Non Surgical Protocol for Treatment of Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Clementini, Principal Investigator, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mucositis non surgical
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Peri-implant Mucositis
Keywords: peri-implant mucositis; non surgical therapy; laser; air powder
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechanical debridement with curettes (Sham Comparator): mechanical debridement: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments
  Interventions: Procedure: Mechanical debridement with curettes
- Er:YAG laser (Experimental): Er:YAG laser treatment will be provided on the implant/abutment surface.
  Interventions: Procedure: Er:YAG laser
- Air Powder (Active Comparator): an Air-Powder treatment will be provided on the implant/abutment surface.
  Interventions: Procedure: Air Powder

INTERVENTIONS:
Procedure: Mechanical debridement with curettes — mechanical debridement: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments
  Arms: Mechanical debridement with curettes
Procedure: Er:YAG laser — mechanical debridement: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments. Furthermore, an Er:YAG laser will be used for the implant surface decontamination.
  Arms: Er:YAG laser
Procedure: Air Powder — mechanical debridement: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments. Furthermore, an Air-Powder treatment will be provided on the implant/abutment surface.
  Arms: Air Powder

SUMMARY:
Peri-implant mucositis is an important disease entity as a result of its high prevalence and the lack of a standard mode of therapy.

Non-surgical therapy of peri-implant mucositis appears to be partially effective in resolving the disease. In several cases, however, only limited improvements have been reported in the main clinical parameters (bleeding partial resolution and presence of pocket at follow-up visits) and there is a clear tendency to relapse of the disease.

In these cases it is therefore recommended to consider adjunctive therapies. Numerous approaches have been used for implant surface decontamination including mechanical, chemical and treatments by means of air-powder or laser.

The aim of the present randomized controlled clinical trial will be to assess the efficacy in improving clinical parameters of two further methods of implant surface decontamination (Er:YAG laser or air-abrasive device) after mechanical cleaning during non surgical treatment of peri-implant mucositis.

DETAILED DESCRIPTION:
Peri-implant mucositis, defined as an inflammatory lesion of the surrounding peri-implant tissues without loss of supporting bone, is an important disease entity as a result of its high prevalence and the lack of a standard mode of therapy. Although the current epidemiological data are limited, peri-implant mucositis affects 43% of the subjects.

Numerous approaches have been used for implant surface decontamination, including mechanical, chemical and laser treatments. Using conventional mechanical means, eradication of pathogens on implant surfaces with threads and often with rough surface structures is difficult. Treatment models, such as debridement, effectively used to treat teeth with periodontitis, cannot be used in the same way on rough threaded implant surfaces. The implant rough surface structure also provides the bacteria with ''protected areas'', inaccessible to conventional mechanical removal.

A treatment protocol that may offer an advantage over traditional mechanical treatment includes the use of laser therapy. Data have shown that treatments with Er:YAG lasers have a bactericidal effect. Er:YAG laser treatment can debride the implant surface effectively and safely. Slightly better clinical results in terms of bleeding on probing and clinical attachment level have been reported by Er:YAG laser treatment as compared with traditional non-surgical mechanical debridement with curettes and chlorhexidine.

The air abrasive method for the removal of bacterial plaque on tooth surfaces has also been used in the treatment of mucositis, demonstrating no relevant adverse effects. Until recently, air-polishing devices have used a slurry of water and sodium bicarbonate (NaHCO3) and pressurized air/water. A less abrasive method using an aminoacid glycine has been proven to be effective in removing bacterial biofilm structures in deep periodontal pockets and safe by not causing emphysema. Moreover the use of a glycine-based powder does not seem to cause titanium implant surface changes.

The aim of the present randomized controlled clinical trial will be to assess the efficacy in improving clinical parameters of two further methods of implant surface decontamination (Er:YAG laser or air-abrasive device) after mechanical cleaning during non surgical treatment of mucositis.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least one screw-type titanium implant exhibiting bleeding and/or suppuration on probing combined without progressive radiographic bone loss (compared to crestal bone levels at the time of placement of the reconstruction)or <3mm bone level
* single tooth and bridgework restorations without overhangings
* no evidence of occlusal overload (i.e. occlusal contacts revealed appropriate adjustment)
* implant function time ≥ 1 year

Exclusion Criteria:

* Patients with uncontrolled diabetes
* patients with osteoporosis or under bisphosphonate medication,
* pregnant or lactating women,
* patients with a history of radiotherapy to the head and neck region
* patients with incapability to perform basal oral hygiene measures due to physical or mental disorders
* hollow implants
* implant mobility
* implants at which no position could be identified where proper probing measurements could be performed;
* previous surgical treatment of the peri-implantitis lesions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing changes | baseline, 1, 3, 6 months
  changes of bleeding on probing, evaluated as present if bleeding will be evident within 30 s after probing, or absent, if no bleeding will be noticed within 30 s after probing

SECONDARY OUTCOMES:
probing pocket depth changes | baseline, 1, 3, 6 months
  changes in probing pocket depth, measured from the mucosal margin to the bottom of the probable pocket
mucosal recession changes | baseline, 1, 3, 6 months
  changes in mucosal recession, measured from the mucosal margin to the restoration margin or implant neck
clinical attachment level changes | baseline, 1, 3, 6 months
  changes in clinical attachment level, measured from the restoration margin or implant neck to the bottom of the probable pocket at six aspects per implant (mesio-vestibular, mid-vestibular, disto-vestibular, mesio-oral, mid-oral, and disto-oral.
complete disease resolution (percentage) | 6 months
  At the implant level, the level of disease resolution was defined as complete when BoP was = 0 out of six sites per implant

CONTACTS AND LOCATIONS:
Overall Officials: Massimo De Sanctis, Study Chair — Università Vita-Salute San Raffaele
Locations (1):
- Università Vita-Salute San Raffaele, Milan, Italy